CLINICAL TRIAL: NCT06095388
Title: Phase I/II Study of Weekly Infusions of JR-441 in Patients With Mucopolysaccharidosis Type IIIA
Brief Title: Phase I/II Study of JR-441 in Patients With Mucopolysaccharidosis Type IIIA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: JCR Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JR-441-101
Record Dates: First submitted 2023-09-13; First posted 2023-10-23 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Mucopolysaccharidosis III-A
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JR-441 low dose (Experimental)
  Interventions: Drug: JR-441
- JR-441 medium dose (Experimental)
  Interventions: Drug: JR-441
- JR-441 high dose (Experimental)
  Interventions: Drug: JR-441

INTERVENTIONS:
Drug: JR-441 — IV infusion
  Other Names: posnafusp alfa
  Arms: JR-441 low dose
Drug: JR-441 — IV infusion
  Other Names: posnafusp alfa
  Arms: JR-441 medium dose
Drug: JR-441 — IV infusion
  Other Names: posnafusp alfa
  Arms: JR-441 high dose

SUMMARY:
A Phase I/ II, open-label, randomized, 2-arm study, designed to evaluate the safety and explore efficacy of the study drug in development for the treatment of MPS IIIA patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronological age of ≥1 year and ≤18 years.
* Confirmed diagnosis of MPS IIIA.
* Body weight ≥ 10 kg.

Exclusion Criteria:

* Prior experience to gene therapy or HSCT with successful engraftment.
* Past use of another investigational drug or product in last 4 months or 5 half-lives (whichever is longer) before signing ICF.
* Current participation in a clinical trial or past participation (within 30 days of enrolment into this study) in a study involving invasive procedures.
* Past use of Genistein or Kineret (anakinra) within 4 months before signing ICF.
* Serious drug allergy or hypersensitivity.
* Contraindication for lumbar puncture or MRI.
* History of bleeding disorder or current use of medications that, in the opinion of the investigator, place them at risk of bleeding following lumbar puncture.

The above information is not intended to contain all considerations relevant to a patient's potential participation in this clinical trial.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the tolerability of JR-441 in MPSIIIA patients | up to 5 years (multiple visits)
  Adverse events will be reported and graded, laboratory tests will be conducted and vital signs will be monitored
To assess the safety of JR-441 in MPSIII-A patients | up to 5 years (multiple visits)
  Number and severity of infusion-associated reactions, including anaphylaxis

SECONDARY OUTCOMES:
Plasma drug concentration | up to 5 years (multiple visits)
Plasma PK parameters | up to 5 years (multiple visits)
Change from baseline in heparan sulfate levels in cerebrospinal fluid (CSF), serum and urine | up to 5 years (multiple visits)
Change from baseline in cognitive function | up to 5 years (multiple visits)
  Bayley Scales of Infant and Toddler Development, Third Edition (BSID-III) and/or Kaufman Assessment Battery for Children, Second Edition (KABC-II)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany